CLINICAL TRIAL: NCT05510219
Title: Safety Analysis of Intravenous Rapid Infusion of Obinutuzumab in Patients With B-cell
Brief Title: Safety Analysis of Intravenous Rapid Infusion of Obinutuzumab in Patients With B-cell Non-Hodgkin's Lymphoma in China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-169
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Obinutuzumab; Rapid Infusion; Intravenous Infusion Reaction

STUDY DESIGN:
Intervention Model Description: This study was a prospective, single-arm, open-label, phase IV clinical trial that included patients with B-cell non-Hodgkin's lymphoma who visited the Department of Hematology, Jiangsu Provincial People's Hospital . All patients were treated with the standard infusion regimen of obinutuzumab in cycle 1, and for patients who did not develop severe infusion-related reactions (IRRs) in cycle 1, a rapid 90-min obinutuzumab infusion regimen was used from cycle 2 onward while recording any occurrence of infusion reactions in different treatment cycles.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravenous rapid infusion of obinutuzumab (Experimental): Patients with B-cell non-Hodgkin's lymphoma were treated with the standard infusion regimen of obinutuzumab in cycle 1, and for patients who did not develop severe infusion-related reactions in cycle 1, a rapid 90-min obinutuzumab infusion regimen was used from cycle 2 onward while recording any occurrence of infusion reactions in different treatment cycles.
  Interventions: Drug: intravenous rapid infusion of obinutuzumab

INTERVENTIONS:
Drug: intravenous rapid infusion of obinutuzumab — This study was a prospective, single-arm, open-label, phase IV clinical trial that included patients with B-cell non-Hodgkin's lymphoma who visited the Department of Hematology, Jiangsu Provincial People's Hospital. All patients were treated with the standard infusion regimen of obinutuzumab in cycle 1, and for patients who did not develop severe infusion-related reactions (IRRs) in cycle 1, a rapid 90-min obinutuzumab infusion regimen was used from cycle 2 onward while recording any occurrence of infusion reactions in different treatment cycles.

SUMMARY:
This study aimed to analyze the safety of 90-min intravenous rapid infusion of obinutuzumab in patients with B-cell non-Hodgkin's lymphoma and to provide evidence for the applicability of rapid infusion regimens in chemotherapy in China.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of B-cell lymphoma and with indications for obinutuzumab treatment
* No significant organ damage
* ECOG score of 0-2;
* Life expectancy ≥ 6 months
* Informed consent

Exclusion Criteria:

* Pregnant or lactating
* Serologically tested positive for human immunodeficiency virus or hepatitis B virus infection but had not received treatment
* Severe hepatic or renal insufficiency
* Severe cardiovascular disease.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline infusion-related reactions at cycle 6 | at the end of cycle 6(each cycle is 21~28 days)
  The severity of an IRR was graded according to the Common Terminology Criteria for Adverse Events ver 5.0 published by the National Cancer Institute

CONTACTS AND LOCATIONS:
Overall Officials: JianYong Li, doctor, Study Director — Jiangsu Provincial People's Hospital
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China